CLINICAL TRIAL: NCT05474131
Title: Pediatric Out-of-hospital Cardiopulmonary Arrest, Current Status of Out-of-hospital Management, Predictive Factors of Mortality, Physicians' Attitudes, Training Perspectives : a Multicentric Retrospective Study.
Brief Title: Pediatric Out-of-hospital Cardiopulmonary Arrest
Acronym: Ped-CPA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-07Obs-CHRMT
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Pediatric; Cardiac Arrest; Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational and retrospective study is to determine the predictive factors of in-hospital mortality following an out-of-hospital cardiopulmonary arrest (CPA) in the population under 18 years old. Data are collected from telephone calls and medical regulation records processed by the health call center of 2 french departments between January 1, 2019, and March 15, 2022. The medical records of the included patients will also be reread in order to obtain the patient's status at 30 days after the CPA.

Detailed description:

The literature reports numerous works evaluating the epidemiological characteristics of pediatric out-of-hospital cardiorespiratory arrest. An improvement in survival has been reported in the case of resuscitation guided by the operator in medical regulation before the arrival of the emergency services. Indeed, the regulation phase at the 15 center in France is of fundamental importance. Recent evolutions, notably with the creation of specific call-taking professions, show the importance attached to improving practices.

The population concerned is characterized by children under 18 years of age, victims of an extra-hospital cardiorespiratory arrest. It is a retrospective study over three years and three months, multicentric, from the emergency service (SAMU) 57 and 69.

The primary endpoint was the all-cause mortality at thirty days of the admission.

The case report form (CRF) will collect the main aspects of telephone management at the 15 centers, out-of-hospital management by the emergency teams, and the personal characteristics of the emergency physicians and out-of-hospital responders (gender, age, family situation, etc.). The medical management in the emergency department and the first stages of in-hospital management will also be analyzed. The patients included who are still alive will receive a notification of non-objection by mail.

ELIGIBILITY:
Inclusion Criteria:

* child under 17 years old
* and call for cardiac arrest or cardiac arrest detected on call

Exclusion Criteria:

* non-real cardiac arrest

Ages: 1 Day to 17 Years | Sex: All
Age Groups: Child
Study Population: population under 18 years old, with out-of-hospital cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
death from any cause within thirty days of admission | at day 30
  The vital status at Day 30 will be systematically sought.

SECONDARY OUTCOMES:
Resuscitation in pre-hospital care during the listening of the sound tapes of the SAMU | at day 1
  The resumption of a spontaneous cardiac activity will be sought during the listening of the sound tapes of the SAMU

CONTACTS AND LOCATIONS:
Overall Officials: Laure ABENSUR VUILLAUME, PhD, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France